CLINICAL TRIAL: NCT02719119
Title: Trial of Monthly Versus Bi-weekly Endoscopic Variceal Ligation for the Prevention of Esophageal Variceal Rebleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: monthly versus bi-weekly EVL
Record Dates: First submitted 2016-03-19; First posted 2016-03-25 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Esophageal and Gastric Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- monthly EVL (Experimental): Elective band ligation was applied after premedication with hyoscine-N-butylbromide (20 mg intramuscularly). A multiband ligator and video endoscopes were utilized. Ligation was initiated at or slightly below the bleeding point. During each treatment session, each varix was ligated with one or two elastic bands. Variceal obliteration success was when all varices disappeared or residual varices were too small to be ligated further. Once esophageal varices were obliterated, surveillance endoscopy was performed every 3 months for 1 year and then every 6 months to check for recurrent varices. Patients in this group will underwent endoscopic variceal ligation monthly.
  Interventions: Procedure: monthly Endoscopic Variceal Ligation (EVL)
- bi-weekly EVL (Experimental): Elective band ligation was applied after premedication with hyoscine-N-butylbromide (20 mg intramuscularly). A multiband ligator and video endoscopes were utilized. Ligation was initiated at or slightly below the bleeding point. During each treatment session, each varix was ligated with one or two elastic bands. Variceal obliteration success was when all varices disappeared or residual varices were too small to be ligated further. Once esophageal varices were obliterated, surveillance endoscopy was performed every 3 months for 1 year and then every 6 months to check for recurrent varices. Patients in this group will underwent endoscopic variceal ligation bi-weekly.
  Interventions: Procedure: bi-weekly Endoscopic Variceal Ligation (EVL)

INTERVENTIONS:
Procedure: monthly Endoscopic Variceal Ligation (EVL) — Patients in this group will underwent endoscopic variceal ligation monthly.
  Arms: monthly EVL
Procedure: bi-weekly Endoscopic Variceal Ligation (EVL) — Patients in this group will underwent endoscopic variceal ligation bi-weekly.
  Arms: bi-weekly EVL

SUMMARY:
Many physicians suggest repeating EVL every 1-2 weeks until esophageal varices are obliterated to prevent variceal rebleeding， however, the evidences supporting the efficacy of EVL intervals of 1-2 weeks are insufficient.This randomized controlled study was conducted in order to compare the long-term results of EVL when performed at two different results from monthly and bi-weekly treatments.

DETAILED DESCRIPTION:
Endoscopic variceal ligation (EVL) is a safe and simple procedure now being used on a widening scale. A lot of patients who undergo endoscopic treatment for esophageal varices eventually require additional treatment for recurrent varices. Many physicians suggest repeating EVL every 1-2 weeks until esophageal varices are obliterated to prevent variceal rebleeding， however, the evidences supporting the efficacy of EVL intervals of 1-2 weeks are insufficient.This randomized controlled study was conducted in order to compare the long-term results of EVL when performed at two different results from monthly and bi-weekly treatments.

ELIGIBILITY:
Inclusion Criteria:

1. acute or recent bleeding from esophageal varices;
2. portal hypertension caused by cirrhosis;
3. age between 18 and 80 yr.

Exclusion Criteria:

1. history of endoscopic, pharmacological, interventional or surgical treatment of esophageal varices;
2. presence of liver failure with a serum total bilirubin concentration greater than 3 mg/dL;
3. presence of hepatocellular carcinoma or other malignancy;
4. an association with a cerebral vascular accident, uremia, acute coronary syndrome, or other severe illness;
5. history of gastric variceal bleeding;
6. encephalopathy of stage II or worse;
7. failure to control initial variceal bleeding;
8. death within 48 h of admission;
9. refusal to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
variceal rebleeding rate | 2 years

SECONDARY OUTCOMES:
gastrointestinal rebleeding rate | 2 years
variceal obliteration rate | 2 years
number of sessions required to abstain variceal obliteration | 2 years
adverse events | 2 years
mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: li yang, MD, Study Chair — department of gastroenterology
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided